CLINICAL TRIAL: NCT00580567
Title: Impulsivity in Pathological Gambling: A Cross Sectional Analysis on Tests of Impulsivity Between Pathological Gamblers and a Non-pathological Control Group.
Brief Title: Impulsivity in Pathological Gambling
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Timothy Fong MD, Associate Professor of Psychiatry, National Institute on Drug Abuse (NIDA)
Other Study IDs: PA-00-004; K23DA019522 (NIH); PA-00-004
Record Dates: First submitted 2007-12-20; First posted 2007-12-24 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Pathological Gambling
Keywords: Impulsivity; Gambling; Pathological Gamblers; Problem Gamblers; Non-Pathological Gamblers; Risk-taking; Inhibition; Gambling Severity
MeSH Terms: conditions — Gambling; Impulsive Behavior; Risk-Taking; Inhibition, Psychological

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Pathological Gamblers
- 2: Non-Pathological Gamblers

SUMMARY:
The purpose of the this study is to compare pathological gamblers versus non-pathological gamblers using tests that measure different components of impulsivity. We aim to invite a total of 120 individuals to participate in this study.

Impulsivity has been described as the cognitive inability to delay gratification, a failure to inhibit behavioral action or acting without forethought about consequences. Impulsivity has also been seen as a personality trait characterized by risk-taking or sensation seeking behavior. Pathological gamblers demonstrate aspects of impulsivity; they act without thinking, have difficult inhibiting urges to gamble and desire immediate gratification. The goal of this project is to clarify which components of impulsivity are associated with pathological gambling. Non-treatment seeking, pathological gamblers and controls will be recruited from the community and local casinos. Each participant will be administered a battery of tests that represent different operational definitions of impulsivity.

DETAILED DESCRIPTION:
Personality traits of impulsivity will be measured with the Barrett Impulsiveness Scale and the NEO Personality Inventory-Revised. Behavioral components of impulsivity will be tested through delay and probability discounting tasks. Finally, measures of frontotemporal functioning are also included in a neuropsychology and neurocognitive battery. Recent studies have shown that these areas of the brain function differently in pathological gamblers; thus, the following neuropsychology/neurocognitive tests have been included: Attention/Information Processing Speed (via Simple Reaction Time Task and Continuous Performance Task), Episodic Memory (via Hopkins Verbal Learning Test-Revised and Brief Visuospatial Memory Test), Executive/Frontal Lobe Measures (via Wechsler Memory Scale-III, Choice Reaction Time Task, Working Memory Task (N-back), Probabilistic Reversal Learning Task, and Stop-Signal Task). Between group comparisons on this battery of impulsivity tests will be made to clarify which components of impulsivity are associated with pathological gambling. Secondly, within-group analyses will be performed to correlate impulsivity to gambling severity. Lastly, an exploratory analysis of subtyping pathological gamblers by performances on tasks of impulsivity and types of gambling will be conducted.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Pathological Gamblers:

* 18 years or older
* Be able to speak, read and write in English
* Current diagnosis of pathological gambling (using DSM-IV criteria)
* South Oaks Gambling Screen (SOGS) score of 5 or above during screening
* Recent gambling activity -- at least once within one week prior to enrollment.
* Voluntarily given informed consent and signed the informed consent document.
* Not currently seeking treatment for gambling

Inclusion Criteria For Control Participants:

* 18 years or older
* Be able to speak, read and write in English
* South Oaks Gambling Screen (SOGS) score of 5 or less during screening
* Voluntarily given informed consent and signed the informed consent document
* Does not meet diagnosis of pathological gambling by DSM-IV criteria
* Not currently seeking treatment for gambling

Exclusion Criteria:

Exclusion Criteria for all participants:

* Current treatment for pathological gambling, excluding involvement with Gamblers Anonymous
* Ongoing medication for any psychiatric disorders, including anti-psychotics, antidepressants, mood stabilizers, anxiolytics or sedative/hypnotics.
* Dependence by DSM-IV criteria on any psychoactive substance, excluding caffeine or nicotine
* Presence of clinically unstable medical disorders that could harm the subject if not treated immediately.
* Presence of any neurological or psychiatric disorders (as assessed by the SCID or MINI and BDI-II) that would require immediate treatment.
* Test positive urine toxicology for illicit drugs prior to enrollment
* Hamilton Depression Scale score of >17

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community Sample
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2007-03; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Barratt Impusivity Scale | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Timothy W. Fong, M.D., Principal Investigator — UCLA Gambling Studies Program
Locations (1):
- UCLA Neuropsychiatric Institute, Los Angeles, California, United States

REFERENCES:
- See also: UCLA Gambling Studies Program — http://www.uclagamblingprogram.org/